CLINICAL TRIAL: NCT02569060
Title: Feeding America Intervention Trial for Health--Diabetes Mellitus
Acronym: FAITH-DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Feeding America (Other); Laura and John Arnold Foundation (Other); Urban Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A125548
Record Dates: First submitted 2015-10-02; First posted 2015-10-06 (Estimated); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Diabetes Mellitus
Keywords: diabetes mellitus; community intervention; intervention; randomized; dietary intervention; self-management support; food bank
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate Intervention (Experimental): Participants randomized to the Intervention Arm will immediately begin a four-component intervention.
  1. Testing and monitoring of blood glucose levels
  2. Referral to and/or coordination with primary care provider
  3. Diabetes-appropriate food packages
  4. Diabetes self-management education and support
  Interventions: Other: Testing and Monitoring of Blood Glucose Levels; Other: Primary care coordination; Other: Diabetes-appropriate food packages; Behavioral: Diabetes self-management education
- Waitlist Control (Active Comparator): Participants randomized to the Waitlist Control arm will receive no intervention for six months, after which time they will begin a modified, four-component intervention.
  1. Testing and monitoring of blood glucose levels
  2. Referral to and/or coordination with primary care provider
  3. Diabetes-appropriate food packages
  4. Limited diabetes self-management education and support
  Interventions: Other: Testing and Monitoring of Blood Glucose Levels; Other: Primary care coordination; Other: Diabetes-appropriate food packages; Behavioral: Diabetes self-management education

INTERVENTIONS:
Other: Testing and Monitoring of Blood Glucose Levels — Point-of-care testing of HbA1c levels at the food pantry at approximately 3 month intervals
Other: Primary care coordination — Referral to a local primary care provider, if none currently exists. Coordination of care with primary care provider.
Other: Diabetes-appropriate food packages — Food (perishable and non-perishable) appropriate for diabetes self-management available for pick-up at the food pantry twice monthly.
Behavioral: Diabetes self-management education — Education materials drawn from evidence-based practice and adapted from existing diabetes education curricula to be flexible to individual, community, and site variations. The Immediate Intervention Arm receives more robust diabetes self-management education (with group education visits) than the Waitlist Control Arm.

SUMMARY:
The Feeding America Intervention Trial for Health-Diabetes Mellitus (FAITH-DM) is a randomized, controlled study of the implementation of a diabetes intervention in food pantry settings.

DETAILED DESCRIPTION:
For adults with diabetes mellitus, diabetes self-management education (DSME) is critical to achieving long-term control of blood sugar levels (glycemic control) and preventing diabetes-associated complications. This education is often difficult to access for highly vulnerable and marginalized adults in the United States. Furthermore, foods for a diabetic diet are often out of reach for food insecure households. The purpose of this study is to determine the extent to which food banks and food pantries can help reach this population with effective DSME, food, and access to primary health care. The investigators' primary outcome of interest is HbA1c improvement in the intervention group compared to a wait-listed control group of food pantry clients living with uncontrolled type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Food pantry client at one of three participating food banks: Alameda County Community Food Bank (Oakland, CA), Gleaners Community Food Bank of Southeastern Michigan (Detroit, MI), Houston Food Bank, (Houston, TX)
* Type II diabetes mellitus with HbA1c ≥ 7.5% using food bank point-of-care testing
* Reliable mode of contact (either phone or address)
* English or Spanish verbal fluency
* 18 years of age or older
* Intent to remain in the study area for at least the next 12 months
* Willingness to participate in intervention

Exclusion Criteria:

* Type 1 diabetes
* Pregnant or less than 6 weeks post-partum
* Cognitively impaired: dementia, mental illness, or active substance abuse severe enough to interfere with administration of the survey or participation in the intervention
* Household member already enrolled in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 568 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline HbA1c at 6 Months | 6 months
  Point-of-care HbA1c testing with the PTS Diagnostics A1CNow®+ System

SECONDARY OUTCOMES:
Change from Baseline Dietary Intake | 6 months and 12 months
  Brief fruit & vegetable dietary screener
Change from Baseline Health Care Utilization | 6 months and 12 months
  Communication with primary care provider requesting dates of service, service levels, and diagnosis codes
Change from Baseline Diabetes Distress | 6 months and 12 months
  Self-reported distress as assessed by the 2-item emotional burden sub-score of the Diabetes Distress Scale
Change from Baseline Hypoglycemic events | 6 months and 12 months
  Self-reported hypoglycemic events over the previous 4 weeks, both any events and number of events, and self-reported severe hypoglycemic episodes, both any events and number of events
Change from Baseline Depressive symptoms | 6 months and 12 months
  PHQ-8 (a subset of PHQ-9 scores without assessment of suicidality)
Change from Baseline Medication Adherence | 6 months and 12 months
  Morisky Medication Adherence Scale (4 items)
Food vs medicine trade-offs | 6 months and 12 months
  Three self-reported questions
Change from Baseline Food security status | 6 months and 12 months
  6-item version of the USDA's Core Food Security Survey Module
Change from Baseline Food stability | 6 months and 12 months
  Two items assessing adequacy of food resources to last the entire month

OTHER OUTCOMES:
Change from Baseline Diabetes Self-Efficacy | 6 months and 12 months
  8-item scale of diabetes-specific self-efficacy
Change from Baseline Diabetes Self-Care | 6 months and 12 months
  Self-reported assessment of 5 self-care behaviors: medications, exercise, diet, blood sugar monitoring, and foot care

CONTACTS AND LOCATIONS:
Overall Officials: Hilary K Seligman, MD MAS, Principal Investigator — University of California, San Francisco
Locations (4):
- United States (4):
  - Alameda County Community Food Bank, Oakland, California
  - University of California San Francisco, San Francisco, California
  - Gleaners Community Food Bank of Southeastern Michigan, Detroit, Michigan
  - Houston Food Bank, Houston, Texas

REFERENCES:
- [Derived] Seligman HK, Levi R, Ridberg R, Smith M, Hills N, Waxman E. Impact of Enhanced Food Pantry Services on Food Security among Adults with Diabetes Using a Crossover Study Design. Curr Dev Nutr. 2022 Feb 10;6(4):nzac021. doi: 10.1093/cdn/nzac021. eCollection 2022 Apr. PMID 35415385
- [Derived] Smith M, Rosenmoss S, Seligman HK. Point-of-Care Hemoglobin A1C Testing System in Community Settings: Challenges, Opportunities, and Measurement Characteristics. Prog Community Health Partnersh. 2020;14(3):327-335. doi: 10.1353/cpr.2020.0038. PMID 33416608
- [Derived] Seligman HK, Smith M, Rosenmoss S, Marshall MB, Waxman E. Comprehensive Diabetes Self-Management Support From Food Banks: A Randomized Controlled Trial. Am J Public Health. 2018 Sep;108(9):1227-1234. doi: 10.2105/AJPH.2018.304528. Epub 2018 Jul 19. PMID 30024798

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-05): https://cdn.clinicaltrials.gov/large-docs/60/NCT02569060/Prot_SAP_000.pdf